CLINICAL TRIAL: NCT03788304
Title: High Flow Nasal Cannula Versus Non-invasive Ventilation in Prevention of Escalation to Invasive Mechanical Ventilation in Patients With Acute Hypoxemic Respiratory Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Entsar Hsanen Mohamed, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: High flow nasal cannula
Record Dates: First submitted 2018-12-20; First posted 2018-12-27 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: patients with will be randomly enrolled to either non invasive group or HFNC group and improvement and patient satisfaction will be assessed
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the participant , care provider , the investigator nor the outcome assessor will select patients in both groups , see results of other patients till the end of the study or informed by literature opinion in this intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non invasive ventilation (Active Comparator): Respiratory assistance is provided by a NIV either Puritan Bennet 840 , Engström Carestation or Hamilton-G5 , will be used for conventional non-invasive ventilation via an oronasal mask. Settings will be adjusted based on the clinical assessment of the respiratory therapist . Initial setting includes: -
  * Positive End Expiratory Pressure (PEEP): 5 cmH2O.
  * Pressure support (PS): 12-20 cmH2O.
  * FiO2 will be adjusted to achieve a SpO2 at least 95%
  Interventions: Device: non-invasive ventilation
- High flow nasal cannula (Experimental): High flow nasal cannula consists of an apparatus that allows adjustable FiO2 from 21 to 100% and delivers a modified gas flow up to 60 l/ min .
  will be set with: -
  * Temperature at 37°C or 34°C
  * Flow rate 30: 50 L/min.
  * FiO2 will be adjusted to achieve a SpO2 at least 95%
  Interventions: Device: high flow nasal cannula

INTERVENTIONS:
Device: non-invasive ventilation — conventional NIV
  Arms: Non invasive ventilation
Device: high flow nasal cannula — HFNC ventilation
  Arms: High flow nasal cannula

SUMMARY:
Oxygen therapy is first-line treatment in the management of acute respiratory failure (ARF). Different oxygen devices have become available over recent decades, such as low-flow systems (nasal cannula, simple facemask, non-rebreathing reservoir mask) and high-flow systems (Venturi mask) . Since the 90's, non-invasive ventilation (NIV) has been largely used with strong level of evidence in cardiogenic pulmonary edema and chronic obstructive pulmonary disease (COPD) exacerbation. NIV improves gas exchange and reduces inspiratory effort through positive pressure. However, good tolerance to NIV is sometimes difficult to achieve due to frequent leaks around the mask, possibly leading to patient-ventilator asynchrony and even to intubation . High-flow nasal oxygen therapy (HFNO) is an innovative high-flow system that allows for delivering up to 60 liters\ min of heated and fully humidified gas with a FIO2 ranging between 21% and 100% . It is a new method of respiratory support in adults that has been used in neonatal ARF for some years. The reason this study is necessary is because, even though NIV has been demonstrated to prevent endotracheal intubation (and its associated complications) in a broad range of ARF patients, HFNC has been proposed to have the same effect as NIV while being easier tolerated, more physiological , allowing patients to continue to talk, eat and drink through mouth while on HFNC

DETAILED DESCRIPTION:
Oxygen therapy is the first-line treatment in management of acute respiratory failure (ARF). Different oxygen delivery devices have become available over recent decades, either low-flow systems (nasal cannula, simple facemask, non-rebreathing reservoir mask) or high-flow systems (Venturi mask) . The choice of a specific device in management of ARF is based on the severity of hypoxemia, the underlying mechanisms, the patient's breathing pattern and tolerance .

Critically ill patients often require high-flow devices to meet their oxygen needs . Tachypneic patients with ARF, have a peak inspiratory flow rate that is usually high and often exceeds the oxygen flow delivered by the traditional oxygen devices . Using conventional devices, oxygen flow is limited to no more than 15 L/min. Meanwhile, the required inspiratory flow for patients with respiratory failure varies widely in a range from 30 to120 L/min. The difference between patient inspiratory flow and delivered flow is large with conventional oxygen devices leading to patient discomfort . Moreover; high respiratory rate can generate significant entrainment of room air in the mask and dilution of the inspired oxygen with an insufficient oxygen concentration. The suboptimal humidification of the inhaled oxygen provided by standard bubble humidifiers and the limited and unknown inspiratory oxygen fraction (FIO2) delivery are additional drawbacks of these devices .

Since the 90's, noninvasive ventilation (NIV) has been largely used with strong level of evidence in cardiogenic pulmonary edema and chronic obstructive pulmonary disease (COPD) exacerbation. NIV improves gas exchange and reduces inspiratory effort through positive pressure. However, good tolerance to NIV is sometimes difficult to achieve due to frequent leaks around the mask, possibly leading to patient-ventilator asynchrony and even to intubation. It may have other deleterious effects such as delayed intubation by masking signs of respiratory distress, or barotrauma by the high tidal volume potentially generated under positive pressure .

To ensure good results, an appropriate interface is more important than the ventilation mode . Oronasal masks, nasal masks, and hoods are most commonly used for NIV. Oronasal masks are usually tried first because they ensure the effects of NIV better than other interfaces. Unfortunately, it is not comfortable, and many patients find it hard to tolerate. It is also associated with a relatively high incidence of air leakage. Also, skin lesions at the nose induced by long-term use of this device may result in frequent treatment interruptions and discontinuation.

High-flow nasal oxygen therapy (HFNO) is an innovative high-flow system that allows for delivering up to 60 liters/ min of heated and fully humidified gas with a FIO2 ranging between 21% and 100% [.

* HFNO delivery systems: main technical characteristics: - The administration of HFNO requires the following: high pressure sources of oxygen and air, an air-oxygen blender or a high-flow 'Venturi' system (which permits delivery of an accurate FIO2 between 21% and 100%), a humidifying and heating system for conditioning the gas to optimal temperature (37 ºC) and humidity (44mg H2O/ liters), a sterile water reservoir, a non-condensing circuitry, and an interface . The two most widely marketed HFNO systems are the Precision Flow by Vapotherm and Optiflow by Fisher & Pykel Healthcare Ltd.
* Physiological effects of HFNC: - Gas from an air/oxygen blender that can generate a total flow of up to 60 L/min is heated and humidified with an active humidifier and subsequently delivered through a heated circuit. High flow of adequately heated and humidified gas is considered to have a number of physiological effects

  1. Washout of nasopharyngeal dead space: Washout of upper airway dead space from the delivery of a large amount of oxygen can improve the efficiency of ventilation and enhance oxygen delivery . HFNC is the only noninvasive respiratory support that does not increase dead space. With an oxygen mask, especially at low flow, carbon dioxide is rebreathed .
  2. Warming and humidification of secretions: Warming of inspired oxygen and heating it to core temperature is more effective at high flow rates (typically >40 L/minute) than low flow rates. Thus, HFNC is better at heating and humidifying inspired oxygen than conventional high-flow systems such as Venturi masks or nonrebreathers (flow rate typically 10 to 15 L/minute) or low-flow systems (flow rates typically <10 L/minute) . Increased humidification results in increased water content in mucous, which can facilitate secretion removal and may also decrease the work of breathing and avoid airway desiccation and epithelial injury
  3. Continuous positive airway pressure (CPAP) effect: Several studies in adults have shown that, similar to infants and neonates, HFNC increases nasopharyngeal airway pressure that peaks at the end of expiration (ie, "PEEP effect") . This "PEEP effect" can potentially unload auto-PEEP, decrease work of breathing, and enhance oxygenation in patients with alveolar filling diseases such as congestive heart failure or acute respiratory distress syndrome (ARDS). As flow increases, nasopharyngeal pressure increases (ie, a dose effect) . The CPAP effect is greatest with the mouth closed. In general, every increase of 10 L/minute of flow yields approximately 0.7 cm H2O of airway pressure when the mouth is closed and 0.35 cm of H2O when the mouth is open.
  4. Small pliable nasal prongs: HFNC nasal prongs are generally soft and pliable. Consequently, several studies have reported improved patient comfort with HFNC when compared with conventional low-flow oxygen delivered through nasal cannula or high-flow oxygen delivered through a face mask .
  5. High flow rates: High flow rates result in minimal entrainment of room air when HFNC is used; this results in more accurate delivery of oxygen. Patients in respiratory distress generate high inspiratory flow rates that exceed flow rates of standard oxygen equipment, resulting in entrainment of room air and a reduction in the delivery of the set FIO2. The rate of flow in HFNC generally exceeds that of the patient, entraining very little room air and resulting in an FIO2 that is more reliably delivered . High flow rates have also been shown to result in an improved breathing pattern by increasing tidal volume and decreasing respiratory rate .
  6. Reduction of work of breathing: The HFNO system may significantly reduce the energy requirement (metabolic work) associated with gas conditioning. By providing high gas flows, HFNO reduces the resistance of the upper airway and then decreases the resistive breathing effort .

ELIGIBILITY:
Inclusion Criteria:

* Participants admitted to the RICU with acute hypoxemic respiratory failure requiring NIV support with the following criteria:

  1. RR> 25 breath/minute
  2. Use of accessory muscles of respiration, paradoxical breathing, thoracoabdominal asynchrony.
  3. Hypoxemia evidenced by PaO2 / FiO2 ratio <300

Exclusion Criteria:

Patients who have any of the following:

I. Indication for emergency endotracheal intubation. II. HR <50 beat\minute with decreased level of consciousness III. Persistent hemodynamic instability with

* Systolic blood pressure <90 mmHg after infusing a bolus of crystalloid solution at a dose of 30 ml / kg
* life-threatening arrhythmia. IV. Undrained pneumothorax or Pneumothorax with persistent air leak. V. Extensive facial trauma or burn VI. Refusal to participate. VII. Usual long-term treatment with NIV for chronic disease VIII. Altered mental status with decreased consciousness and/or evidence of inability to understand .

IX. Tracheotomy or other upper airway disorders X. Active upper gastrointestinal bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Endotracheal intubation rate. | one week
  needs escalation to invasive mechanical ventilation

SECONDARY OUTCOMES:
In hospital mortality. | one week
  death
length of hospital stay | one week
  hospital coast
duration of ICU stay | one week
  icu occupancy
duration of intervention | one week
  need ventilatory support
development of complications | one week
  due to devices

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed F Adam, lecturer, Principal Investigator — Assiut University; Manal A El-Khawaga, lecturer, Principal Investigator — Assiut University
Locations (1):
- Assiut University hospital, Asyut, Egypt

REFERENCES:
- [Background] 1-Renda, T., Corrado, A., Iskandar, G., et al. High-flow nasal oxygen therapy in intensive care and anaesthesia . British journal of anaesthesia 2018 , 120(1), 18-27 2-Kallstrom TJ. AARC clinical practice guideline: oxygen therapy for adults in the acute care facility: 2002 revision and update. Respir Care 2002; 47: 717-20. 3-O'Driscoll BR, Howard LS, Davison AG, on behalf of the British Thoracic Society. BTS guideline for emergency oxygen use in adult patients. Thorax 2008; 63: 1-68. 4-Sim MA, Dean P, Kinsella J, et al. Performance of oxygen delivery devices when the breathing pattern of respiratory failure is simulated. Anaesthesia 2008; 63: 938-40 5-Nishimura, M. High-flow nasal cannula oxygen therapy in adults: physiological benefits, indication, clinical benefits, and adverse effects. Respiratory Care 2016, 61(4), 529-541.